CLINICAL TRIAL: NCT00088413
Title: An Open Label Pilot Study to Evaluate the Safety and Tolerability of PANVAC-V (Vaccinia) and PANVAC-F (Fowlpox) in Combination With Sargramostim in Adults With Metastatic Carcinoma
Brief Title: PANVAC-V and PANVAC-F Vaccines Plus Sargramostim to Treat Advanced Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, James Gulley, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 040246; 04-C-0246; NCT00091000 (obsolete NCT alias)
Record Dates: First submitted 2004-07-23; First posted 2004-07-26 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Adenocarcinoma; Colorectal Cancer; Ovarian Cancer; Breast Cancer
Keywords: CEA; Vaccine; Immunotherapy; MUC-1; Cancer; Adenocarcinoma; Metastatic Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma; Colorectal Neoplasms; Ovarian Neoplasms; Breast Neoplasms; Neoplasms | interventions — sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All Cohorts: Colorectal, Non-Colorectal, Breast, and Ovarian (Experimental): All cohorts receive the same intervention (Cohort 1: Colorectal arm, non-colorectal cancers; Cohort 2: breast cancer; Cohort 3: ovarian cancers)
  Interventions: Biological: PANVAC-V; Biological: PANVAC-F; Drug: Sargramostim (GM-CSF, Leukine)

INTERVENTIONS:
Biological: PANVAC-V — Patients receive 2 x 10(8) pfu PANVAC-V (vaccinia) subcutaneously on Day 1.
Biological: PANVAC-F — Patients receive 1 x 10(9) pfu PANVAC-F (fowlpox) or about days 15, 29, and 43 then every month for 12 doses then every 3 months until disease progression or toxicity.
Drug: Sargramostim (GM-CSF, Leukine) — 100g sargramostim will be given subcutaneously at the site of the vaccination on each vaccination day and for three consecutive days thereafter.
  Other Names: Granulocyte-macrophage colony-stimulating factor

SUMMARY:
Background:

* Many cancers produce two proteins, carcinoembryonic antigen (CEA) and mucin-1 (MUC-1).
* The PANVAC-V (PANVAC vaccinia) priming vaccine and PANVAC-F (PANVAC fowlpox) boosting vaccine contain human genes that cause production of CEA and MUC-1, which can be used as a target for the immune system to attack the cancer. The vaccines also contain genes that cause production of other proteins that enhance immune activity.
* Sargramostim is a protein that boosts the immune system.

Objectives:

* To evaluate the safety and effectiveness of PANVAC-V and PANVAC-F in patients with advanced cancer.
* To document the immune response to the vaccines and any anti-tumor responses that may occur.

Eligibility: Patients 18 years of age and older with advanced cancer whose tumors produce CEA or MUC-1 protein

Design:

* This trial has three cohorts: the first cohort includes 10 patients with advanced colorectal cancer and 10 to 15 patients with any advanced non-colorectal cancer that produces either EA or mitochondrial Ca2+ uniporter 1 (MCU-1); the second cohort includes 12 patients with advanced breast cancer and the third cohort includes 14 patients with advanced ovarian cancer.
* All patients receive PANVAC-V on study day 1, followed by PANVAC-F on days 15, 29 and 43 then every 28 days for up to 12 vaccines followed by every 3 months until disease progression or toxicity. The vaccines are given by injection under the skin. Sargramostim is injected at the vaccination site on the day of each vaccination and for the next 3 days following vaccination.
* Patients whose scans show that their disease has progressed, but who are otherwise clinically stable may revert back to monthly injections.
* Patients undergo apheresis to collect white blood cells (lymphocytes) on day 1 and day 71 of the study to measure the immune response to the treatment. Blood is collected through a needle placed in one arm and directed through a cell separator machine where the lymphocytes are extracted. The rest of the blood components are returned to the patient through the same needle.
* Patients are monitored with frequent blood tests and periodic imaging tests (scans) to monitor for safety and the response to treatment.

DETAILED DESCRIPTION:
Background:

* Carcinoembryonic antigen (CEA) and mucin-1 (MUC-1) are overexpressed in multiple adenocarcinomas.
* Pox viral vectors can induce a strong immune response to CEA and MUC-1.
* The use of agonist epitopes within the tumor associated antigen (TAA) can induce a better immune response than native peptides and have been associated with clinical responses
* Heterologous prime and boost regimens are superior in terms of generalizing immune responses; and this may translate into improved clinical responses
* The use of granulocyte-macrophage colony-stimulating factor (GM-CSF) does not add significant toxicity and in pre-clinical models is essential for induction for optimal immune responses.
* It is possible by using vectors directed against TAA that there may be additive or synergistic immune responses and this may be important in overcoming antigenic escape variance
* Evidence of clinical benefit has been noted in some patients treated with this vaccine

Objectives:

* For colorectal cancer and non-colorectal cancer Cohort: To evaluate the safety and tolerability of the vaccine.
* For the Ovarian Cancer and Breast Cancer Cohorts: To evaluate clinical response to the vaccine.

Eligibility:

* In the first cohort (colorectal and non-colorectal cancer), histologically confirmed adenocarcinoma that is CEA or MUC-1 positive described as metastatic disease (measurable or evaluable) or metastatic disease documented by biopsy but not evaluable by imaging (e.g. small volume peritoneal disease)
* For the ovarian and breast cancer cohorts, patients must have evaluable disease
* Normal organ function, Eastern Cooperative Oncology Group (ECOG) 0-1

Design:

* This is a non-randomized three cohort, pilot trial of pox viral vaccines that contain the transgenes for CEA and MUC-1 (both with modified human leukocyte antigen A2 (HLA-A2) agonist epitopes) as well as 3 human T-cell costimulatory molecules, B7-1, ICAM-1 (CD54), and LFA-3 (CD58) [PANVAC(TM)-V (vaccinia) and PANVAC(TM)-F (fowlpox)] in patients with metastatic carcinoma that express CEA or MUC-1 antigen.
* The first cohort will enroll 10 patients with metastatic colorectal adenocarcinoma and 10-15 patients with any metastatic non-colorectal carcinoma that expresses either CEA or MUC-1. .
* The second cohort will enroll 12 patients with metastatic breast carcinoma and 14 patients with metastatic ovarian carcinoma.
* All patients will receive the same vaccines on the same schedule. PANVAC(TM)-V (vaccinia) subcutaneously (s.c.) scheduled on day 1, followed by PANVAC(TM)-F (fowlpox) s.c. scheduled on days 15, 29, and 43 then every 28 days for up to 12 vaccines followed by every 3 months until disease progression or toxicity.
* Sargramostim (100 micro g) will be given at the site of the vaccination (PANVAC-V and PANVAC-F) on each vaccination day and for three consecutive days thereafter.
* Patients who have radiographic evidence of progressive disease, but who are otherwise clinically stable may revert back to monthly vaccinations.

ELIGIBILITY:
* INCLUSION CRITERIA:

A. Histologically confirmed carcinoma that for patients in the first cohort (colorectal and non-colorectal cancer) is carcinoembryonic antigen (CEA) or mucin-1 (MUC-1) positive. Tumor that has been shown to express CEA or MUC-1 (greater than or equal to 20 % of cells) by immunohistochemical techniques or patients that have had an elevated serum CEA (greater than 5 microgram/L) at any point during their disease course. For patients in the ovarian and breast cancer cohorts, as greater than 95% of these express MUC-1 or CEA, we will not require staining prior to coming onto trial.

B. Patients must have completed at least one fluorouracil (5-FU) containing chemotherapy regimen (e.g. 5-FU/leucovorin (LV) with or without either irinotecan or oxaliplatin) for the colorectal cancer arm, or either failed or not be a candidate for therapy of proven efficacy for non-colorectal, breast, or ovarian cancer.

C. 18 years of age or greater.

D. All patients enrolled on the colorectal/non-colorectal cohort with colorectal adenocarcinoma cohort must be human leukocyte antigen A2 (HLA-A2) positive.

E. At least 10 patients enrolled on the colorectal/non-colorectal cohort with non-colorectal adenocarcinoma cohort must be HLA-A2 positive.

F. Patients in the breast cohort and the ovarian cohorts are not required to be HLA-A2 positive.

G. For the colorectal and non-colorectal cancer cohort, patients will be required to have: metastatic disease (measurable or evaluable), metastatic disease documented by biopsy but not evaluable by imaging (e.g. small volume peritoneal disease), and patients with surgically resected metastatic disease at high risk of relapse. For the ovarian cohort and the breast cancer cohort, patients will be required to have evaluable disease.

H. Able to understand and give informed consent.

I. Able to avoid close household contact (close household contacts are those who share housing or have close physical contact) for at least three weeks after recombinant vaccinia vaccination with persons with active or a history of eczema or other eczematoid skin disorders; those with other acute, chronic or exfoliative skin conditions (e.g., atopic dermatitis, burns, impetigo, varicella zoster, severe acne, or other open rashes or wounds) until condition resolves; pregnant or nursing women; children 3 years of age and under; and immunodeficient or immunosuppressed persons (by disease or therapy), including human immunodeficiency virus (HIV) infection.

J. Eastern Oncology Cooperative Group (ECOG) performance status of 0 - 1.

K. Serum creatinine not above the institution limits of normal, and aspartate aminotransferase (AST) less than or equal to twice the upper limits of normal OR creatinine clearance on a 24 hour urine collection of greater than or equal to 60 mL/min.

L. Total bilirubin within the institution limits of normal OR patients with Gilbert's syndrome, a total bilirubin less than or equal to 3.0

M. Recovered completely from any reversible toxicity associated with recent therapy. Typically this is 3-4 weeks for patients who most recently received cytotoxic therapy except for the nitrosoureas and mitomycin C for which 6 weeks is needed for recovery.

N. Hematological eligibility parameters (within 16 days of starting therapy):

* Granulocyte count greater than or equal to 1,500/mm(3)
* Platelet count greater than or equal to 100,000/mm(3)
* Hemoglobin (Hgb) greater than or equal to 10 Gm/dL

O. Prior immune therapy with related vaccinia and fowlpox vaccines or antigen-specific peptides is allowed.

P. Men and women must agree to use effective birth control or abstinence during and for a period of 4 months after the last vaccination therapy.

Q. Patients with prostate cancer must continue to receive gonadotropin-releasing hormone (GnRH) agonist therapy (unless orchiectomy has been done).

R. Patients should appear clinically stable (in the opinion of the principal investigator) to complete the full 3 month course of vaccination with an anticipated survival of 6 months or longer.

EXCLUSION CRITERIA:

A. Patients should have no evidence of being immunocompromised as listed below.

* Human immunodeficiency virus positivity due to the potential for decreased tolerance and risk for severe side effects
* Active autoimmune diseases requiring treatment or a history of autoimmune disease that might be stimulated by vaccine treatment. This requirement is due to the potential risks of exacerbating autoimmunity. Patients with endocrine disease that is controlled by replacement therapy including thyroid disease and adrenal disease and vitiligo may be enrolled.

B. Concurrent use of systemic steroids, except for physiologic doses for systemic steroid replacement or local (topical, nasal, or inhaled) steroid use. Limited doses systemic steroids to prevent intravenous (IV) contrast, allergic reaction, or anaphylaxis (in patients who have known contrast allergies) are allowed.

C. History of allergy or untoward reaction to prior vaccination with vaccinia virus.

D. Pregnant or breast-feeding women.

E. Altered immune function, including immunodeficiency or history of immunodeficiency; eczema; history of eczema, or other eczematoid skin disorders; or those with acute, chronic or exfoliative skin conditions (e.g. atopic dermatitis, burns, impetigo, varicella zoster, severe acne, or other open rashes or wounds).

F. Serious intercurrent medical illness which would interfere with the ability of the patient to carry out the treatment program, including, but not limited to, inflammatory bowel disease, Crohn's disease, ulcerative colitis, or active diverticulitis

G. Patients with a history of cardiomyopathy or symptomatic congestive heart failure (unless stable on treatment), symptomatic arrhythmia not controlled by medication. Unstable atherosclerotic heart disease (e.g. unstable angina) who require active intervention and history of myocardial infarction or embolic stroke within the past 6 months.

H. Clinically active brain metastasis, or a history of encephalitis, multiple sclerosis, or seizures within the last year (from seizure disorder or brain metastasis).

I. Medical conditions, which, in the opinion of the investigators would jeopardize the patient or the integrity of the data obtained.

J. Concurrent chemotherapy; an exception to this is to allow for patients with breast cancer who are receiving trastuzumab, to continue therapy with trastuzumab while receiving the vaccine treatment.

K. Serious hypersensitivity reaction to egg products.

L. Clinically significant cardiomyopathy requiring treatment.

M. Chronic hepatitis infection, including B and C, because of potential immune impairment.

N. Although topical steroids are allowed, steroid eye drop are contraindicated.

O. Cardiac complications, including recent myocardial infarction or cerebrovascular accident within one year, and/or unstable or uncontrolled angina.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2004-07-21 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James L Gulley, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Madan RA, Bilusic M, Heery C, Schlom J, Gulley JL. Clinical evaluation of TRICOM vector therapeutic cancer vaccines. Semin Oncol. 2012 Jun;39(3):296-304. doi: 10.1053/j.seminoncol.2012.02.010. PMID 22595052
- [Background] Madan RA, Arlen PM, Gulley JL. PANVAC-VF: poxviral-based vaccine therapy targeting CEA and MUC1 in carcinoma. Expert Opin Biol Ther. 2007 Apr;7(4):543-54. doi: 10.1517/14712598.7.4.543. PMID 17373905
- [Result] Mohebtash M, Tsang KY, Madan RA, Huen NY, Poole DJ, Jochems C, Jones J, Ferrara T, Heery CR, Arlen PM, Steinberg SM, Pazdur M, Rauckhorst M, Jones EC, Dahut WL, Schlom J, Gulley JL. A pilot study of MUC-1/CEA/TRICOM poxviral-based vaccine in patients with metastatic breast and ovarian cancer. Clin Cancer Res. 2011 Nov 15;17(22):7164-73. doi: 10.1158/1078-0432.CCR-11-0649. Epub 2011 Nov 8. PMID 22068656
- [Result] Gulley JL, Arlen PM, Tsang KY, Yokokawa J, Palena C, Poole DJ, Remondo C, Cereda V, Jones JL, Pazdur MP, Higgins JP, Hodge JW, Steinberg SM, Kotz H, Dahut WL, Schlom J. Pilot study of vaccination with recombinant CEA-MUC-1-TRICOM poxviral-based vaccines in patients with metastatic carcinoma. Clin Cancer Res. 2008 May 15;14(10):3060-9. doi: 10.1158/1078-0432.CCR-08-0126. PMID 18483372
- [Derived] Gorodetska I, Samusieva A, Lahuta T, Ponomarova O, Socha O, Kozeretska I. Exploring New Frontiers: Alternative Breast Cancer Treatments Through Glycocalyx Research. Breast J. 2025 May 22;2025:9952727. doi: 10.1155/tbj/9952727. eCollection 2025. PMID 40443562

RESULTS

PARTICIPANT FLOW:
Groups:
- Colorectal Cancer Cohort: Patients with histologically confirmed measurable or evaluable metastatic colorectal cancer or patients with surgically resected metastatic disease at high risk for recurrence who had completed at least one 5-fluorouracil/(5-FU) containing chemotherapy regimen (e.g., 5-fluorouracil/leucovorin (5-FU/LV) with or without either irinotecan or oxaliplatin or patients that have had an elevated serum CEA (>5 ugg/L) at any point during their disease course who have failed or not a candidate for standard therapy.
- Non-Colorectal Cancer Cohort: Patients with histologically confirmed measurable or evaluable metastatic non-colorectal cancer or patients with surgically resected metastatic disease at high risk for recurrence who had completed at least one 5-fluorouracil/(5-FU) containing chemotherapy regimen (e.g., 5-fluorouracil/leucovorin (5-FU/LV) with or without either irinotecan or oxaliplatin or patients that have had an elevated serum CEA (>5 ugg/L) at any point during their disease course who have failed or not a candidate for standard therapy.
- Breast Cohort: Patients with evaluable, metastatic breast cancer who have failed or not a candidate for standard therapy.
- Ovarian Cohort: Patients with evaluable, metastatic ovarian cancer who have failed or not a candidate for standard therapy.
Period: Overall Study
Arm/Group | Colorectal Cancer Cohort | Non-Colorectal Cancer Cohort | Breast Cohort | Ovarian Cohort
Started | 10 | 15 | 12 | 14
Completed | 0 | 0 | 0 | 0
Not Completed | 10 | 15 | 12 | 14
Not completed — Limited supply of trmt drug (PANVAC-f) | 0 | 0 | 1 | 0
Not completed — Adverse Events/Side Effects | 0 | 1 | 1 | 0
Not completed — Refused trmt Off-study per pt wishes | 0 | 1 | 1 | 0
Not completed — Off study due to missing a vaccine dose | 1 | 0 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0
Not completed — Progressive disease | 9 | 11 | 8 | 14
Not completed — Other | 0 | 1 | 0 | 0
Not completed — Patient unevaluable due to adverse event | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Colorectal Cancer Cohort: Patients with histologically confirmed measurable or evaluable colorectal cancer or patients with surgically resected metastatic disease at high risk for recurrence who had completed at least one 5-fluorouracil/(5-FU) containing chemotherapy regimen (e.g., 5-fluorouracil/leucovorin (5-FU/LV) with or without either irinotecan or oxaliplatin or patients that have had an elevated serum CEA (>5 ugg/L) at any point during their disease course who have failed or not a candidate for standard therapy.
- Total: Total of all reporting groups
Arm/Group | Colorectal Cancer Cohort | Non-Colorectal Cancer Cohort | Breast Cohort | Ovarian Cohort | Total
Number analyzed (Participants) | 10 | 15 | 12 | 14 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 12 | 10 | 12 | 42
  >=65 years | 2 | 3 | 2 | 2 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (12.2) | 57.6 (7.91) | 56.5 (11.8) | 54.8 (9.0) | 55.6 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 13 | 12 | 14 | 43
  Male | 6 | 2 | 0 | 0 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 9 | 15 | 12 | 14 | 50
  Asian | 0 | 1 | 1 | 0 | 2
  Black or African-American | 0 | 1 | 1 | 0 | 2
  White | 10 | 12 | 0 | 0 | 22
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 15 | 12 | 14 | 51
Number of Participants with Eastern Cooperative Oncology Group (ECOG) Performance Status Grade 0-1 [Count of Participants; unit: Participants] — Grade 0 is normal activity. Fully active, able to carry on all pre-disease performance without restriction. Grade 1 is symptoms, but ambulatory. Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature (e.g. light housework, office work).
  Participants
    Grade 0 | 4 | 5 | 2 | 5 | 16
    Grade 1 | 6 | 10 | 10 | 9 | 35
Number of Participants with Prior Therapy [Count of Participants; unit: Participants]
  No prior chemotherapy | 0 | 0 | 1 | 0 | 1
  Chemotherapy (1 regimen) | 2 | 5 | 1 | 1 | 9
  Chemotherapy (2 regimens) | 3 | 6 | 2 | 1 | 12
  Chemotherapy (≥3 regimens) | 5 | 4 | 8 | 12 | 29
  Radiation | 2 | 3 | 8 | 0 | 13
Number of Participants with a Primary Tumor [Count of Participants; unit: Participants]
  Colorectal | 10 | 0 | 0 | 0 | 10
  Gastric | 0 | 3 | 0 | 0 | 3
  Pancreatic | 0 | 2 | 0 | 0 | 2
  Appendiceal | 0 | 2 | 0 | 0 | 2
  Esophageal adenocarcinoma | 0 | 1 | 0 | 0 | 1
  Ovarian | 0 | 3 | 0 | 14 | 17
  Breast | 0 | 2 | 12 | 0 | 14
  Lung | 0 | 2 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Responses (CRs), Partial Responses (PRs,) Stable Disease and Progressive Disease in the Ovarian Cancer and Breast Cancer Cohorts
Description: Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete Response is disappearance of all clinical and laboratory signs and symptoms of disease for a minimum of 4 weeks during which no new lesions may appear. Partial Response is a minimum of 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter. Stable disease is neither sufficient shrinkage to qualify for partial response nor progressive disease, taking as reference the smallest sum longest diameter since the treatment started. Progressive disease is a minimum of 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of one or more new measurable lesions.
Time Frame: Approximately 6 months while on trial
Measure: Count of Participants; unit: Participants
Groups:
- Breast Cancer Cohort: Patients with evaluable, metastatic breast cancer who have failed or not a candidate for standard therapy.
- Ovarian Cancer Cohort: Patients with evaluable, metastatic ovarian cancer who have failed or not a candidate for standard therapy.
Arm/Group | Breast Cancer Cohort | Ovarian Cancer Cohort
Number analyzed (Participants) | 12 | 14
Participants
  Complete Response | 1 | 0
  Partial Response | 0 | 0
  Stable Disease | 4 | 3
  Progressive Disease | 7 | 11

2. Primary Outcome: Percentage of Vaccines Associated With Grade 1 and Grade 2 Adverse Events Related to Vaccine in the Colorectal Cancer and Non-Colorectal Cancer Arm/Group
Description: Grade 1 (mild) and Grade 2 (moderate) adverse events were assessed by the Common Terminology Criteria in Adverse Events (CTCAE) v3.0 if reported prior to August 1, 2010 and CTCAE v4.0 if reported after. A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Approximately 6 months while on trial
Population: The colorectal and non-colorectal cohorts received the same treatment on the same schedule, had no immune dysfunction at baseline and are biologically equivalent. For rare events in small cohorts, a better estimate of the true event rate is determined by grouping similar patients and is consistent with the peer-reviewed clinical paper.
Measure: Number; unit: Percentage of vaccines
Units Other Than Participants: Vaccines administered
Groups:
- Colorectal Cancer and Non-Colorectal Cancer Cohort: Patients with histologically confirmed measurable or evaluable metastatic colorectal cancer, non-colorectal cancer or patients with surgically resected metastatic disease at high risk for recurrence who had completed at least one 5-fluorouracil/(5-FU) containing chemotherapy regimen (e.g., 5-fluorouracil/leucovorin (5-FU/LV) with or without either irinotecan or oxaliplatin or patients that have had an elevated serum CEA (>5 ugg/L) at any point during their disease course who have failed or not a candidate for standard therapy.
Arm/Group | Colorectal Cancer and Non-Colorectal Cancer Cohort
Number analyzed (Participants) | 25
Number analyzed (Vaccines administered) | 180
Percentage of vaccines
  Injection-site reaction | 88
  Fatigue | 5
  Fever | 3
  Hemoglobin/Anemia | 1
  Hypoalbuminemia | 1
  Alk Phos | 1
  Syncope | 0
  Anorexia | 1
  Vomiting | 1
  Hot flushes/flashes | 1

3. Secondary Outcome: Percentage of Participants With Grade 1 and Grade 2 Adverse Events Possibly, Likely, or Definitely Related to Vaccine in the Breast Cancer and Ovarian Cancer Cohorts
Description: Vaccines were administered to participants and Grade 1 (mild) and Grade 2 (moderate) adverse events were assessed by the Common Terminology Criteria in Adverse Events (CTCAE) v3.0 if reported prior to August 1, 2010 and CTCAE v4.0 if reported after. Common Terminology Criteria in Adverse Events. A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Approximately 2 months while on trial
Population: The breast and ovarian cohorts received the same treatment on the same schedule, had no evidence of immune dysfunction at baseline and are biologically equivalent. For rare events that occur in small trial arms, the true event rate is better determined by grouping similar patients and is consistent with the peer-reviewed clinical paper.
Measure: Number; unit: percentage of participants
Groups:
- Breast Cancer and Ovarian Cancer Cohorts: Patients with evaluable, metastatic breast or ovarian cancer who have failed or not a candidate for standard therapy.
Arm/Group | Breast Cancer and Ovarian Cancer Cohorts
Number analyzed (Participants) | 26
percentage of participants
  Injection-site reaction | 22
  Musculoskeletal pain | 2
  Anemia | 1

4. Secondary Outcome: Number of Participants With Adverse Events Assessed by the Common Terminology Criteria in Adverse Events (CTCAE) v3.0 and v4.0
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE) v3.0 if reported prior to August 1, 2010 and CTCAE v4.0 if reported after. A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date consent signed to date off study, approximately 164 months and 10 days
Population: Pts in these 2 cohorts rec'd the same treatment, have absence of immune dysfunction at baseline and are biologically equivalent. For rare events that occur in small cohorts, a better est. of the true event rate can be determined by grouping the pts in the absence of a biological rationale and is consistent with the peer-reviewed clinical paper.
Measure: Count of Participants; unit: Participants
Groups:
- Colorectal Cancer and Non-Colorectal Cancer Cohort: Patients with histologically confirmed measurable or evaluable metastatic colorectal cancer, non-colorectal cancer, or patients with surgically resected metastatic disease at high risk for recurrence who had completed at least one 5-fluorouracil/(5-FU) containing chemotherapy regimen (e.g., 5-fluorouracil/leucovorin (5-FU/LV) with or without either irinotecan or oxaliplatin or patients that have had an elevated serum CEA (>5 ugg/L) at any point during their disease course who have failed or not a candidate for standard therapy.
- Breast Cancer and Ovarian Cancer Cohort: Patients with evaluable, metastatic breast cancer or ovarian cancer who have failed or not a candidate for standard therapy.
Arm/Group | Colorectal Cancer and Non-Colorectal Cancer Cohort | Breast Cancer and Ovarian Cancer Cohort
Number analyzed (Participants) | 25 | 26
Participants | 25 | 26

5. Secondary Outcome: Number of Participants With an Positive Immune Response to Carcinoembryonic Antigen (CEA) Peptide and/or Protein in the Colorectal Cancer and Non-colorectal Cancer Cohort Post Vaccination
Description: Immune response in human leukocyte antigens (HLA)-A2 positive patients to carcinoembryonic antigen (CEA) was assessed by enzyme-linked immunospot assay (ELISPOT) analysis. A positive immune response was defined as a >2x fold increase in the number of interferon gamma producing cells.
Time Frame: post vaccination (up to Day 84)
Population: Overall number of participants analyzed reflects participants that are HLA-A2 positive.
Measure: Count of Participants; unit: Participants
Arm/Group | Colorectal Cancer Cohort | Non-Colorectal Cancer Cohort
Number analyzed (Participants) | 9 | 9
Participants | 3 | 6

6. Secondary Outcome: Number of Participants With an Positive Immune Response to Carcinoembryonic Antigen (CEA) Peptide and/or Protein in the Breast Cancer and Ovarian Cancer Cohorts Post Vaccination
Description: as for outcome 5
Time Frame: post vaccination (up to Day 84)
Population: Only 3 Breast Cancer and 2 Ovarian Cancer patients had enough blood collected to perform enzyme-linked immunospot (ELISPOT) analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Breast Cancer Cohort | Ovarian Cancer Cohort
Number analyzed (Participants) | 3 | 2
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 164 months and 10 days.
Description: Adverse events were assessed by the Common Terminology Criteria in Adverse Events(CTCAE)*v3.0 if reported prior to August 1, 2010 and CTCAE *v4.0 if reported after.
Groups:
- Colorectal Cancer vs Non-Colorectal Cancer Cohort: Patients with histologically confirmed measurable or evaluable metastatic colorectal cancer or patients with surgically resected metastatic disease at high risk for recurrence who had completed at least one 5-fluorouracil/(5-FU) containing chemotherapy regimen (e.g., 5-fluorouracil/leucovorin (5-FU/LV) with or without either irinotecan or oxaliplatin or patients that have had an elevated serum CEA (>5 ugg/L) at any point during their disease course who have failed or not a candidate for standard therapy.
- Breast and Ovarian Cohorts: Patients with evaluable, metastatic breast or ovarian cancer who have failed or not a candidate for standard therapy.
Arm/Group | Colorectal Cancer vs Non-Colorectal Cancer Cohort | Breast and Ovarian Cohorts
All-Cause Mortality (participants affected / at risk) | 1/25 | 0/26
Serious Adverse Events (participants affected / at risk) | 25/25 | 26/26
Other Adverse Events (participants affected / at risk) | 25/25 | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Colorectal Cancer vs Non-Colorectal Cancer Cohort (N=25) | Breast and Ovarian Cohorts (N=26)
METABOLIC/LABORATORY:: Albumin, serum-low (hypoalbuminemia)*3 (General disorders) | 0 (0) | 1 (2)
Activated partial thromboplastin time prolonged*4 (Investigations) | 0 (0) | 1 (1)
Alanine aminotransferase increased*4 (Investigations) | 0 (0) | 1 (5)
Alkaline phosphatase increased*4 (Investigations) | 0 (0) | 1 (1)
Allergic reaction*4 (Immune system disorders) | 0 (0) | 1 (1)
Allergic rhinitis*4 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Anemia*4 (Blood and lymphatic system disorders) | 0 (0) | 1 (8)
Aspartate aminotransferase increased*4 (Investigations) | 0 (0) | 1 (6)
BLOOD/BONE MARROW:: Hemoglobin*3 (Blood and lymphatic system disorders) | 13 (34) | 8 (14)
BLOOD/BONE MARROW:: Leukocytes (total WBC)*3 (Blood and lymphatic system disorders) | 4 (22) | 1 (3)
BLOOD/BONE MARROW:: Lymphopenia*3 (Blood and lymphatic system disorders) | 2 (6) | 1 (2)
BLOOD/BONE MARROW:: Neutrophils/granulocytes (ANC/AGC)*3 (Blood and lymphatic system disorders) | 5 (13) | 1 (4)
BLOOD/BONE MARROW:: Platelets*3 (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Back pain*4 (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bruising*4 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
CARDIAC ARRHYTHMIA:: Supraventricular and nodal arrhythmia:: Sinus tachycardia*3 (Cardiac disorders) | 0 (0) | 1 (1)
CONSTITUTIONAL SYMPTOMS:: Weight gain*3 (General disorders) | 0 (0) | 1 (1)
CPK increased*4 (Investigations) | 0 (0) | 1 (1)
Creatinine increased*4 (Investigations) | 0 (0) | 1 (1)
Cystitis noninfective*4 (Renal and urinary disorders) | 0 (0) | 1 (1)
DERMATOLOGY/SKIN:: Dermatology/Skin - Other (Allergic reaction-Tape)*3 (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DERMATOLOGY/SKIN:: Dry skin*3 (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
DERMATOLOGY/SKIN:: Injection site reaction/extravasation changes*3 (Skin and subcutaneous tissue disorders) | 0 (0) | 23 (83)
Delirium*4 (Psychiatric disorders) | 0 (0) | 1 (1)
Depression*4 (Psychiatric disorders) | 0 (0) | 1 (1)
Diarrhea*4 (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fall*4 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fever*4 (General disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL:: Anorexia*3 (Gastrointestinal disorders) | 5 (6) | 2 (2)
GASTROINTESTINAL:: Constipation*3 (Gastrointestinal disorders) | 3 (4) | 5 (6)
GASTROINTESTINAL:: Dehydration*3 (Gastrointestinal disorders) | 4 (4) | 1 (1)
GASTROINTESTINAL:: Diarrhea*3 (Gastrointestinal disorders) | 5 (8) | 5 (9)
GASTROINTESTINAL:: Distension/bloating, abdominal*3 (Gastrointestinal disorders) | 2 (2) | 1 (1)
GASTROINTESTINAL:: Dysphagia (difficulty swallowing)*3 (Gastrointestinal disorders) | 2 (2) | 1 (1)
GASTROINTESTINAL:: Heartburn/dyspepsia*3 (Gastrointestinal disorders) | 6 (12) | 2 (3)
GASTROINTESTINAL:: Nausea*3 (Gastrointestinal disorders) | 5 (12) | 10 (13)
GASTROINTESTINAL:: Vomiting*3 (Gastrointestinal disorders) | 5 (9) | 5 (8)
Gingival pain*4 (Gastrointestinal disorders) | 0 (0) | 1 (1)
HEMORRHAGE/BLEEDING:: Hemorrhage, GU:: Urinary NOS*3 (Renal and urinary disorders) | 0 (0) | 1 (1)
HEMORRHAGE/BLEEDING:: Hemorrhage/Bleeding - Other (Spotting)*3 (General disorders) | 0 (0) | 1 (1)
Hallucinations*4 (Psychiatric disorders) | 0 (0) | 1 (1)
Headache*4 (Nervous system disorders) | 0 (0) | 1 (1)
Hyperglycemia*4 (Metabolism and nutrition disorders) | 0 (0) | 1 (5)
Hypernatremia*4 (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperuricemia*4 (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminemia*4 (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Hypocalcemia*4 (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Hypoglycemia*4 (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia*4 (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypomagnesemia*4 (Metabolism and nutrition disorders) | 0 (0) | 1 (4)
Hyponatremia*4 (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypophosphatemia*4 (Metabolism and nutrition disorders) | 0 (0) | 1 (5)
INFECTION:: Infection - Other (Lt. lower leg, redness, swelling, & whelts)*3 (Infections and infestations) | 0 (0) | 1 (1)
INFECTION:: Infection with normal ANC or Grade 1 or 2 neutrophils:: Lung (pneumonia)*3 (Infections and infestations) | 0 (0) | 1 (1)
Injection site reaction*4 (General disorders) | 0 (0) | 1 (4)
Investigations - Other, specify*4 (Investigations) | 0 (0) | 1 (1)
LYMPHATICS:: Edema: limb*3 (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Lipase increased*4 (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased*4 (Investigations) | 0 (0) | 1 (9)
METABOLIC/LABORATORY:: Glucose, serum-low (hypoglycemia)*3 (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
METABOLIC/LABORATORY:: Hemoglobinuria*3 (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
METABOLIC/LABORATORY:: Sodium, serum-high (hypernatremia)*3 (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
MUSCULOSKELETAL/SOFT TISSUE:: Muscle weakness, generalized or specific area (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4) — (not due to neuropathy):: Whole body/generalized*3
NEUROLOGY:: Mood alteration:: Agitation*3 (Nervous system disorders) | 0 (0) | 1 (1)
NEUROLOGY:: Neuropathy: motor*3 (Nervous system disorders) | 0 (0) | 1 (1)
Nasal congestion*4 (Renal and urinary disorders) | 0 (0) | 1 (1)
Neck pain*4 (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nervous system disorders - Other, specify*4 (Nervous system disorders) | 0 (0) | 1 (1)
Neutrophil count decreased*4 (Investigations) | 0 (0) | 1 (1)
Non-cardiac chest pain*4 (General disorders) | 0 (0) | 1 (1)
PAIN:: Pain - Other (Burning sensation waist & tumor area)*3 (General disorders) | 0 (0) | 1 (1)
PAIN:: Pain:: Chest/thorax NOS*3 (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN:: Pain:: Pelvis*3 (Reproductive system and breast disorders) | 0 (0) | 3 (3)
PAIN:: Pain:: Throat/pharynx/larynx*3 (Gastrointestinal disorders) | 0 (0) | 1 (1)
PULMONARY/UPPER RESPIRATORY:: Nasal cavity/paranasal sinus reactions*3 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY/UPPER RESPIRATORY:: Pleural effusion (non-malignant)*3 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pain*4 (General disorders) | 0 (0) | 1 (4)
Peripheral motor neuropathy*4 (Nervous system disorders) | 0 (0) | 1 (1)
Pleural effusion*4 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pruritus*4 (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
SYNDROMES:: Flu-like syndrome*3 (General disorders) | 3 (12) | 18 (35)
Sinus bradycardia*4 (Cardiac disorders) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, specify*4 (Surgical and medical procedures) | 0 (0) | 1 (1)
Vomiting*4 (Gastrointestinal disorders) | 0 (0) | 1 (1)
Weight gain*4 (Investigations) | 0 (0) | 1 (2)
Wound dehiscence*4 (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Wound infection*4 (Infections and infestations) | 0 (0) | 1 (2)
ALLERGY/IMMUNOLOGY:: Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip)*3 (Immune system disorders) | 2 (4) | 4 (6)
CARDIAC ARRHYTHMIA:: Palpitations*3 (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC GENERAL:: Hypotension*3 (Cardiac disorders) | 1 (1) | 0 (0)
COAGULATION:: INR (International Normalized Ratio of prothrombin time)*3 (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
COAGULATION:: PTT (Partial Thromboplastin Time)*3 (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
CONSTITUTIONAL SYMPTOMS:: Constitutional Symptoms - Other (Cold )*3 (General disorders) | 1 (1) | 0 (0)
CONSTITUTIONAL SYMPTOMS:: Fatigue (asthenia, lethargy, malaise)*3 (General disorders) | 13 (24) | 10 (20)
CONSTITUTIONAL SYMPTOMS:: Fever (in the absence of neutropenia, (General disorders) | 10 (14) | 13 (18) — where neutropenia is defined as ANC <1.0 x 10e9/L)*3
CONSTITUTIONAL SYMPTOMS:: Insomnia*3 (General disorders) | 1 (2) | 2 (2)
CONSTITUTIONAL SYMPTOMS:: Rigors/chills*3 (General disorders) | 12 (14) | 3 (4)
CONSTITUTIONAL SYMPTOMS:: Sweating (diaphoresis)*3 (General disorders) | 4 (5) | 2 (4)
CONSTITUTIONAL SYMPTOMS:: Weight loss*3 (General disorders) | 1 (1) | 0 (0)
DEATH:: Death not associated with CTCAE term:: Disease progression NOS*3 (General disorders) | 1 (1) | 1 (1)
DERMATOLOGY/SKIN:: Bruising (in absence of Grade 3 or 4 thrombocytopenia)*3 (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
DERMATOLOGY/SKIN:: Induration/fibrosis (skin and subcutaneous tissue)*3 (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DERMATOLOGY/SKIN:: Injection site reaction/extravasation changes*3 (Skin and subcutaneous tissue disorders) | 25 (146) | 23 (83)
DERMATOLOGY/SKIN:: Nail changes*3 (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5)
DERMATOLOGY/SKIN:: Pruritus/itching*3 (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DERMATOLOGY/SKIN:: Rash/desquamation*3 (Skin and subcutaneous tissue disorders) | 2 (4) | 1 (1)
ENDOCRINE:: Hot flashes/flushes*3 (Endocrine disorders) | 1 (1) | 0 (0)
ENDOCRINE:: Thyroid function, low (hypothyroidism)*3 (Endocrine disorders) | 1 (1) | 0 (0)
GASTROINTESTINAL:: Flatulence*3 (Gastrointestinal disorders) | 2 (2) | 0 (0)
GASTROINTESTINAL:: Gastrointestinal - Other (Partial bowel obstruction)*3 (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL:: Mucositis/stomatitis (functional/symptomatic):: Oral cavity*3 (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROINTESTINAL:: Obstruction, GI:: Small bowel NOS*3 (Gastrointestinal disorders) | 1 (6) | 0 (0)
GASTROINTESTINAL:: Taste alteration (dysgeusia)*3 (Gastrointestinal disorders) | 1 (1) | 0 (0)
HEMORRHAGE/BLEEDING:: Hemorrhage, GI:: Lower GI NOS*3 (Gastrointestinal disorders) | 1 (1) | 0 (0)
HEMORRHAGE/BLEEDING:: Hemorrhage, GI:: Rectum*3 (Gastrointestinal disorders) | 1 (1) | 0 (0)
HEMORRHAGE/BLEEDING:: Hemorrhage, GU:: Bladder*3 (Renal and urinary disorders) | 1 (1) | 0 (0)
HEMORRHAGE/BLEEDING:: Hemorrhage, pulmonary/upper respiratory:: Nose*3 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HEPATOBILIARY/PANCREAS:: Pancreatitis*3 (Hepatobiliary disorders) | 1 (1) | 0 (0)
INFECTION:: Infection with normal ANC or Grade 1 or 2 neutrophils:: Sinus*3 (Infections and infestations) | 2 (2) | 0 (0)
INFECTION:: Infection with normal ANC or Grade 1 or 2 neutrophils:: Urinary tract NOS*3 (Infections and infestations) | 2 (2) | 1 (1)
INFECTION:: Infection with unknown ANC:: Urinary tract NOS*3 (Infections and infestations) | 1 (2) | 0 (0)
INFECTION:: Infection with unknown ANC:: Wound*3 (Infections and infestations) | 1 (1) | 0 (0)
LYMPHATICS:: Lymphatics - Other (Edema-Left ankle)*3 (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
METABOLIC/LABORATORY:: ALT, SGPT (serum glutamic pyruvic transaminase)*3 (Metabolism and nutrition disorders) | 8 (18) | 2 (2)
METABOLIC/LABORATORY:: AST, SGOT(serum glutamic oxaloacetic transaminase)*3 (Metabolism and nutrition disorders) | 7 (12) | 8 (8)
METABOLIC/LABORATORY:: Albumin, serum-low (hypoalbuminemia)*3 (Metabolism and nutrition disorders) | 15 (26) | 20 (25)
METABOLIC/LABORATORY:: Alkaline phosphatase*3 (Metabolism and nutrition disorders) | 8 (10) | 5 (6)
METABOLIC/LABORATORY:: Amylase*3 (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
METABOLIC/LABORATORY:: Bicarbonate, serum-low*3 (Metabolism and nutrition disorders) | 2 (5) | 0 (0)
METABOLIC/LABORATORY:: Bilirubin (hyperbilirubinemia)*3 (Metabolism and nutrition disorders) | 8 (12) | 3 (3)
METABOLIC/LABORATORY:: CPK (creatine phosphokinase)*3 (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
METABOLIC/LABORATORY:: Calcium, serum-high (hypercalcemia)*3 (Metabolism and nutrition disorders) | 5 (7) | 0 (0)
METABOLIC/LABORATORY:: Calcium, serum-low (hypocalcemia)*3 (Metabolism and nutrition disorders) | 5 (7) | 2 (2)
METABOLIC/LABORATORY:: Cholesterol, serum-high (hypercholesteremia)*3 (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
METABOLIC/LABORATORY:: Creatinine*3 (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
METABOLIC/LABORATORY:: GGT (gamma-Glutamyl transpeptidase)*3 (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
METABOLIC/LABORATORY:: Glucose, serum-high (hyperglycemia)*3 (Metabolism and nutrition disorders) | 9 (11) | 5 (5)
METABOLIC/LABORATORY:: Lipase*3 (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
METABOLIC/LABORATORY:: Magnesium, serum-high (hypermagnesemia)*3 (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
METABOLIC/LABORATORY:: Magnesium, serum-low (hypomagnesemia)*3 (Metabolism and nutrition disorders) | 4 (11) | 5 (9)
METABOLIC/LABORATORY:: Phosphate, serum-low (hypophosphatemia)*3 (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
METABOLIC/LABORATORY:: Potassium, serum-high (hyperkalemia)*3 (Metabolism and nutrition disorders) | 2 (3) | 2 (2)
METABOLIC/LABORATORY:: Potassium, serum-low (hypokalemia)*3 (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
METABOLIC/LABORATORY:: Proteinuria*3 (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
METABOLIC/LABORATORY:: Sodium, serum-low (hyponatremia)*3 (Metabolism and nutrition disorders) | 7 (10) | 4 (4)
METABOLIC/LABORATORY:: Uric acid, serum-high (hyperuricemia)*3 (Metabolism and nutrition disorders) | 5 (14) | 2 (2)
NEUROLOGY:: Dizziness*3 (Nervous system disorders) | 5 (8) | 1 (2)
NEUROLOGY:: Mood alteration:: Anxiety*3 (Nervous system disorders) | 2 (2) | 0 (0)
NEUROLOGY:: Mood alteration:: Depression*3 (Nervous system disorders) | 1 (1) | 1 (1)
NEUROLOGY:: Neuropathy: cranial:: CN I Smell*3 (Nervous system disorders) | 1 (1) | 0 (0)
NEUROLOGY:: Neuropathy: cranial:: CN VIII Hearing and balance*3 (Nervous system disorders) | 1 (1) | 0 (0)
NEUROLOGY:: Syncope (fainting)*3 (Nervous system disorders) | 2 (2) | 0 (0)
OCULAR/VISUAL:: Keratitis (corneal inflammation/corneal ulceration)*3 (Eye disorders) | 1 (1) | 0 (0)
OCULAR/VISUAL:: Vision-blurred vision*3 (Eye disorders) | 1 (1) | 0 (0)
PAIN:: Pain:: Abdomen NOS*3 (Gastrointestinal disorders) | 5 (9) | 6 (8)
PAIN:: Pain:: Back*3 (Musculoskeletal and connective tissue disorders) | 10 (11) | 5 (6)
PAIN:: Pain:: Bladder*3 (Renal and urinary disorders) | 1 (1) | 0 (0)
PAIN:: Pain:: Bone*3 (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
PAIN:: Pain:: Chest wall*3 (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
PAIN:: Pain:: Extremity-limb*3 (Musculoskeletal and connective tissue disorders) | 6 (6) | 4 (4)
PAIN:: Pain:: Eye*3 (Eye disorders) | 1 (1) | 1 (1)
PAIN:: Pain:: Head/headache*3 (Nervous system disorders) | 12 (20) | 11 (17)
PAIN:: Pain:: Joint*3 (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0)
PAIN:: Pain:: Muscle*3 (Musculoskeletal and connective tissue disorders) | 12 (20) | 4 (4)
PAIN:: Pain:: Neck*3 (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
PAIN:: Pain:: Oral cavity*3 (Gastrointestinal disorders) | 1 (1) | 0 (0)
PAIN:: Pain:: Pain NOS*3 (General disorders) | 1 (1) | 0 (0)
PAIN:: Pain:: Stomach*3 (Gastrointestinal disorders) | 2 (2) | 1 (1)
PULMONARY/UPPER RESPIRATORY:: Bronchospasm, wheezing*3 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY/UPPER RESPIRATORY:: Cough*3 (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 7 (9)
PULMONARY/UPPER RESPIRATORY:: Dyspnea (shortness of breath)*3 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
RENAL/GENITOURINARY:: Bladder spasms*3 (Renal and urinary disorders) | 1 (2) | 0 (0)
RENAL/GENITOURINARY:: Renal/Genitourinary - Other (Dysuria)*3 (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL/GENITOURINARY:: Urinary frequency/urgency*3 (Renal and urinary disorders) | 2 (2) | 1 (1)
Dermatology/Skin - Other (Mouth sore-lower lip)*3 (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL:: Gastrointestinal - Other (Emesis)*3 (Gastrointestinal disorders) | 1 (1) | 1 (1)
GASTROINTESTINAL:: Gastrointestinal - Other (Erythema Mucosa-Under tongue & hard palate)*3 (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL:: Gastrointestinal - Other (Gastroesophageal reflux disease )*3 (Gastrointestinal disorders) | 0 (0) | 1 (1)
PAIN:: Pain - Other (Right inguinal pain)*3 (General disorders) | 0 (0) | 1 (1)
PAIN:: Pain - Other (Rt. thigh pain)*3 (General disorders) | 0 (0) | 1 (2)
PAIN:: Pain - Other (Sternum pain)*3 (General disorders) | 0 (0) | 1 (1)
PAIN:: Pain - Other (Pain-Upper right quadrant)*3 (General disorders) | 1 (1) | 0 (0)
PAIN:: Pain - Other (Rt. flank)*3 (General disorders) | 1 (1) | 0 (0)
PAIN:: Pain - Other (Rt. ear)*3 (General disorders) | 1 (1) | 0 (0)
PAIN:: Pain - Other (Pain from inserted biliary stents)*3 (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Colorectal Cancer vs Non-Colorectal Cancer Cohort (N=25) | Breast and Ovarian Cohorts (N=26)
ALLERGY/IMMUNOLOGY:: Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip)*3 (Immune system disorders) | 2 (4) | 1 (2)
Activated partial thromboplastin time prolonged*4 (Investigations) | 0 (0) | 4 (6)
Alanine aminotransferase increased*4 (Investigations) | 0 (0) | 1 (1)
Alkaline phosphatase increased*4 (Investigations) | 0 (0) | 1 (1)
Allergic reaction*4 (Immune system disorders) | 0 (0) | 1 (1)
Allergic rhinitis*4 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Anemia*4 (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Aspartate aminotransferase increased*4 (Investigations) | 0 (0) | 1 (6)
BLOOD/BONE MARROW:: Hemoglobin*3 (Blood and lymphatic system disorders) | 13 (34) | 1 (1)
BLOOD/BONE MARROW:: Leukocytes (total WBC)*3 (Blood and lymphatic system disorders) | 4 (22) | 8 (14)
BLOOD/BONE MARROW:: Lymphopenia*3 (Blood and lymphatic system disorders) | 2 (6) | 1 (3)
BLOOD/BONE MARROW:: Neutrophils/granulocytes (ANC/AGC)*3 (Blood and lymphatic system disorders) | 5 (13) | 1 (2)
BLOOD/BONE MARROW:: Platelets*3 (Blood and lymphatic system disorders) | 3 (3) | 1 (4)
Back pain*4 (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Bruising*4 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
CARDIAC ARRHYTHMIA:: Supraventricular and nodal arrhythmia:: Sinus tachycardia*3 (Cardiac disorders) | 0 (0) | 1 (1)
CONSTITUTIONAL SYMPTOMS:: Fatigue (asthenia, lethargy, malaise)*3 (General disorders) | 13 (24) | 1 (1)
CONSTITUTIONAL SYMPTOMS (General disorders) | 0 (0) | 10 (20) — Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L)*3
CONSTITUTIONAL SYMPTOMS:: Insomnia*3 (General disorders) | 1 (2) | 13 (18)
CONSTITUTIONAL SYMPTOMS:: Rigors/chills*3 (General disorders) | 12 (14) | 2 (2)
CONSTITUTIONAL SYMPTOMS:: Sweating (diaphoresis)*3 (General disorders) | 4 (5) | 3 (4)
CONSTITUTIONAL SYMPTOMS:: Weight gain*3 (General disorders) | 0 (0) | 2 (4)
CPK increased*4 (Investigations) | 0 (0) | 1 (1)
Creatinine increased*4 (Investigations) | 0 (0) | 1 (1)
Cystitis noninfective*4 (Renal and urinary disorders) | 0 (0) | 1 (1)
DERMATOLOGY/SKIN:: Dermatology/Skin - Other (Allergic reaction-Tape )*3 (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DERMATOLOGY/SKIN:: Dry skin*3 (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
DERMATOLOGY/SKIN:: Injection site reaction/extravasation changes*3 (Skin and subcutaneous tissue disorders) | 25 (146) | 2 (2)
DERMATOLOGY/SKIN:: Pruritus/itching*3 (Skin and subcutaneous tissue disorders) | 1 (1) | 23 (83)
DERMATOLOGY/SKIN:: Rash/desquamation*3 (Skin and subcutaneous tissue disorders) | 2 (4) | 5 (5)
Delirium*4 (Psychiatric disorders) | 0 (0) | 1 (1)
Depression*4 (Psychiatric disorders) | 0 (0) | 1 (1)
Diarrhea*4 (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fall*4 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fever*4 (General disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL:: Anorexia*3 (Gastrointestinal disorders) | 5 (6) | 1 (1)
GASTROINTESTINAL:: Constipation*3 (Gastrointestinal disorders) | 3 (4) | 2 (2)
GASTROINTESTINAL:: Diarrhea*3 (Gastrointestinal disorders) | 5 (8) | 5 (6)
GASTROINTESTINAL:: Distension/bloating, abdominal*3 (Gastrointestinal disorders) | 2 (2) | 5 (9)
GASTROINTESTINAL:: Dysphagia (difficulty swallowing)*3 (Gastrointestinal disorders) | 2 (2) | 1 (1)
GASTROINTESTINAL:: Heartburn/dyspepsia*3 (Gastrointestinal disorders) | 6 (12) | 4 (4)
GASTROINTESTINAL:: Nausea*3 (Gastrointestinal disorders) | 5 (12) | 2 (3)
GASTROINTESTINAL:: Vomiting*3 (Gastrointestinal disorders) | 5 (9) | 10 (13)
Gingival pain*4 (Gastrointestinal disorders) | 0 (0) | 5 (8)
HEMORRHAGE/BLEEDING:: Hemorrhage, GU:: Urinary NOS*3 (Renal and urinary disorders) | 0 (0) | 1 (1)
HEMORRHAGE/BLEEDING:: Hemorrhage/Bleeding - Other (Spotting )*3 (General disorders) | 0 (0) | 1 (1)
Hallucinations*4 (Psychiatric disorders) | 0 (0) | 1 (1)
Headache*4 (Nervous system disorders) | 0 (0) | 1 (1)
Hyperglycemia*4 (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperuricemia*4 (Metabolism and nutrition disorders) | 0 (0) | 1 (5)
Hypoalbuminemia*4 (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycemia*4 (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypomagnesemia*4 (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphatemia*4 (Metabolism and nutrition disorders) | 0 (0) | 1 (4)
INFECTION:: Infection - Other (Lt. lower leg, redness, swelling & whelts)*3 (Infections and infestations) | 0 (0) | 1 (1)
INFECTION:: Infection with normal ANC or Grade 1 or 2 neutrophils:: Lung (pneumonia)*3 (Infections and infestations) | 0 (0) | 1 (1)
INFECTION:: Infection with normal ANC or Grade 1 or 2 neutrophils:: Urinary tract NOS*3 (Infections and infestations) | 2 (2) | 1 (1)
Injection site reaction*4 (General disorders) | 0 (0) | 1 (1)
LYMPHATICS:: Edema: limb*3 (Blood and lymphatic system disorders) | 2 (2) | 1 (4)
Lipase increased*4 (Infections and infestations) | 0 (0) | 2 (2)
Lymphocyte count decreased*4 (Investigations) | 0 (0) | 1 (1)
METABOLIC/LABORATORY:: ALT, SGPT (serum glutamic pyruvic transaminase)*3 (Metabolism and nutrition disorders) | 8 (18) | 1 (9)
METABOLIC/LABORATORY:: AST, SGOT(serum glutamic oxaloacetic transaminase)*3 (Metabolism and nutrition disorders) | 7 (12) | 2 (2)
METABOLIC/LABORATORY:: Albumin, serum-low (hypoalbuminemia)*3 (Metabolism and nutrition disorders) | 15 (26) | 8 (8)
METABOLIC/LABORATORY:: Alkaline phosphatase*3 (Metabolism and nutrition disorders) | 8 (10) | 20 (25)
METABOLIC/LABORATORY:: Bilirubin (hyperbilirubinemia)*3 (Metabolism and nutrition disorders) | 8 (12) | 5 (6)
METABOLIC/LABORATORY:: CPK (creatine phosphokinase)*3 (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
METABOLIC/LABORATORY:: Calcium, serum-high (hypercalcemia)*3 (Metabolism and nutrition disorders) | 5 (7) | 2 (2)
METABOLIC/LABORATORY:: Calcium, serum-low (hypocalcemia)*3 (Metabolism and nutrition disorders) | 3 (7) | 2 (2)
METABOLIC/LABORATORY:: Cholesterol, serum-high (hypercholesteremia)*3 (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
METABOLIC/LABORATORY:: Glucose, serum-high (hyperglycemia)*3 (Metabolism and nutrition disorders) | 9 (11) | 1 (1)
METABOLIC/LABORATORY:: Glucose, serum-low (hypoglycemia)*3 (Metabolism and nutrition disorders) | 0 (0) | 5 (5)
METABOLIC/LABORATORY:: Hemoglobinuria*3 (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
METABOLIC/LABORATORY:: Magnesium, serum-high (hypermagnesemia)*3 (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
METABOLIC/LABORATORY:: Magnesium, serum-low (hypomagnesemia)*3 (Metabolism and nutrition disorders) | 4 (11) | 1 (1)
METABOLIC/LABORATORY:: Phosphate, serum-low (hypophosphatemia)*3 (Metabolism and nutrition disorders) | 2 (2) | 5 (9)
METABOLIC/LABORATORY:: Potassium, serum-high (hyperkalemia)*3 (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
METABOLIC/LABORATORY:: Potassium, serum-low (hypokalemia)*3 (Metabolism and nutrition disorders) | 2 (3) | 2 (2)
METABOLIC/LABORATORY:: Proteinuria*3 (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
METABOLIC/LABORATORY:: Sodium, serum-high (hypernatremia)*3 (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
METABOLIC/LABORATORY:: Sodium, serum-low (hyponatremia)*3 (Metabolism and nutrition disorders) | 7 (10) | 1 (1)
METABOLIC/LABORATORY:: Uric acid, serum-high (hyperuricemia)*3 (Metabolism and nutrition disorders) | 5 (14) | 4 (4)
MUSCULOSKELETAL/SOFT TISSUE (Metabolism and nutrition disorders) | 0 (0) | 2 (2) — Muscle weakness, generalized or specific area (not due to neuropathy):: Whole body/generalized*3
NEUROLOGY:: Dizziness*3 (Nervous system disorders) | 5 (8) | 3 (4)
NEUROLOGY:: Mood alteration:: Agitation*3 (Nervous system disorders) | 0 (0) | 1 (2)
NEUROLOGY:: Mood alteration:: Depression*3 (Nervous system disorders) | 1 (1) | 1 (1)
NEUROLOGY:: Neuropathy: motor*3 (Nervous system disorders) | 0 (0) | 1 (1)
Nasal congestion*4 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Neck pain*4 (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nervous system disorders - Other, specify*4 (Nervous system disorders) | 0 (0) | 1 (1)
Neutrophil count decreased*4 (Investigations) | 0 (0) | 1 (1)
Non-cardiac chest pain*4 (General disorders) | 0 (0) | 1 (1)
PAIN:: Pain - Other (Burning sensation waist & tumor area)*3 (General disorders) | 0 (0) | 1 (1)
PAIN:: Pain:: Abdomen NOS*3 (Gastrointestinal disorders) | 5 (9) | 3 (5)
PAIN:: Pain:: Back*3 (Musculoskeletal and connective tissue disorders) | 10 (11) | 6 (8)
PAIN:: Pain:: Bone*3 (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (6)
PAIN:: Pain:: Chest wall*3 (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
PAIN:: Pain:: Chest/thorax NOS*3 (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN:: Pain:: Extremity-limb*3 (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (1)
PAIN:: Pain:: Eye*3 (Eye disorders) | 1 (1) | 4 (4)
PAIN:: Pain:: Head/headache*3 (Nervous system disorders) | 12 (20) | 1 (1)
PAIN:: Pain:: Muscle*3 (Musculoskeletal and connective tissue disorders) | 12 (20) | 11 (17)
PAIN:: Pain:: Pelvis*3 (Reproductive system and breast disorders) | 0 (0) | 4 (4)
PAIN:: Pain:: Stomach*3 (Gastrointestinal disorders) | 2 (2) | 3 (3)
PAIN:: Pain:: Throat/pharynx/larynx*3 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY/UPPER RESPIRATORY:: Cough*3 (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 1 (1)
PULMONARY/UPPER RESPIRATORY:: Dyspnea (shortness of breath)*3 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 7 (9)
PULMONARY/UPPER RESPIRATORY:: Nasal cavity/paranasal sinus reactions*3 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pain*4 (General disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy*4 (Nervous system disorders) | 0 (0) | 1 (2)
Pruritus*4 (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
RENAL/GENITOURINARY:: Urinary frequency/urgency*3 (Renal and urinary disorders) | 2 (2) | 1 (1)
SYNDROMES:: Flu-like syndrome*3 (General disorders) | 3 (12) | 1 (1)
Sinus bradycardia*4 (Cardiac disorders) | 0 (0) | 18 (35)
Vomiting*4 (Gastrointestinal disorders) | 0 (0) | 1 (1)
Weight gain*4 (Investigations) | 0 (0) | 1 (1)
Wound dehiscence*4 (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Wound infection*4 (Infections and infestations) | 0 (0) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 1 (1)
CARDIAC ARRHYTHMIA:: Palpitations*3 (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC GENERAL:: Hypotension*3 (Cardiac disorders) | 1 (1) | 0 (0)
COAGULATION:: INR (International Normalized Ratio of prothrombin time)*3 (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
COAGULATION:: PTT (Partial Thromboplastin Time)*3 (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
CONSTITUTIONAL SYMPTOMS:: Constitutional Symptoms - Other (Cold)*3 (General disorders) | 1 (1) | 0 (0)
CONSTITUTIONAL SYMPTOMS:: Fever (in the absence of neutropenia, where neutropenia is defined as ANC (General disorders) | 10 (14) | 0 (0) — <1.0 x 10e9/L)*3
CONSTITUTIONAL SYMPTOMS:: Weight loss*3 (General disorders) | 1 (1) | 0 (0)
DERMATOLOGY/SKIN:: Bruising (in absence of Grade 3 or 4 thrombocytopenia)*3 (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
DERMATOLOGY/SKIN:: Induration/fibrosis (skin and subcutaneous tissue)*3 (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DERMATOLOGY/SKIN:: Nail changes*3 (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
ENDOCRINE:: Hot flashes/flushes*3 (Endocrine disorders) | 1 (1) | 0 (0)
ENDOCRINE:: Thyroid function, low (hypothyroidism)*3 (Endocrine disorders) | 1 (1) | 0 (0)
GASTROINTESTINAL:: Dehydration*3 (Gastrointestinal disorders) | 3 (3) | 0 (0)
GASTROINTESTINAL:: Flatulence*3 (Gastrointestinal disorders) | 2 (2) | 0 (0)
GASTROINTESTINAL:: Mucositis/stomatitis (functional/symptomatic):: Oral cavity*3 (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROINTESTINAL:: Obstruction, GI:: Small bowel NOS*3 (Gastrointestinal disorders) | 1 (2) | 0 (0)
GASTROINTESTINAL:: Taste alteration (dysgeusia)*3 (Gastrointestinal disorders) | 1 (1) | 0 (0)
HEMORRHAGE/BLEEDING:: Hemorrhage, GI:: Lower GI NOS*3 (Gastrointestinal disorders) | 1 (1) | 0 (0)
HEMORRHAGE/BLEEDING:: Hemorrhage, GI:: Rectum*3 (Gastrointestinal disorders) | 1 (1) | 0 (0)
HEMORRHAGE/BLEEDING:: Hemorrhage, GU:: Bladder*3 (Renal and urinary disorders) | 1 (1) | 0 (0)
HEMORRHAGE/BLEEDING:: Hemorrhage, pulmonary/upper respiratory:: Nose*3 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
INFECTION:: Infection with normal ANC or Grade 1 or 2 neutrophils:: Sinus*3 (Infections and infestations) | 2 (2) | 0 (0)
INFECTION:: Infection with unknown ANC:: Urinary tract NOS*3 (Infections and infestations) | 1 (2) | 0 (0)
LYMPHATICS:: Lymphatics - Other (Edema-left ankle)*3 (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
METABOLIC/LABORATORY:: Amylase*3 (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
METABOLIC/LABORATORY:: Bicarbonate, serum-low*3 (Metabolism and nutrition disorders) | 2 (5) | 0 (0)
METABOLIC/LABORATORY:: Creatinine*3 (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
METABOLIC/LABORATORY:: GGT (gamma-Glutamyl transpeptidase)*3 (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
METABOLIC/LABORATORY:: Lipase*3 (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
NEUROLOGY:: Mood alteration:: Anxiety*3 (Nervous system disorders) | 2 (2) | 0 (0)
NEUROLOGY:: Neuropathy: cranial:: CN I Smell*3 (Nervous system disorders) | 1 (1) | 0 (0)
NEUROLOGY:: Neuropathy: cranial:: CN VIII Hearing and balance*3 (Nervous system disorders) | 1 (1) | 0 (0)
NEUROLOGY:: Syncope (fainting)*3 (Nervous system disorders) | 2 (2) | 0 (0)
OCULAR/VISUAL:: Keratitis (corneal inflammation/corneal ulceration)*3 (Eye disorders) | 1 (1) | 0 (0)
OCULAR/VISUAL:: Vision-blurred vision*3 (Eye disorders) | 1 (1) | 0 (0)
PAIN:: Pain - Other (Pain-upper right quadrant)*3 (General disorders) | 1 (1) | 0 (0)
PAIN:: Pain:: Bladder*3 (Renal and urinary disorders) | 1 (1) | 0 (0)
PAIN:: Pain:: Joint*3 (General disorders) | 4 (5) | 0 (0)
PAIN:: Pain:: Neck*3 (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
PAIN:: Pain:: Oral cavity*3 (Gastrointestinal disorders) | 1 (1) | 0 (0)
PAIN:: Pain:: Pain NOS*3 (General disorders) | 1 (1) | 0 (0)
PULMONARY/UPPER RESPIRATORY:: Bronchospasm, wheezing*3 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RENAL/GENITOURINARY:: Bladder spasms*3 (Renal and urinary disorders) | 1 (2) | 0 (0)
RENAL/GENITOURINARY:: Renal/Genitourinary - Other (Dysuria)*3 (Renal and urinary disorders) | 1 (1) | 0 (0)
DERMATOLOGY/SKIN:: Dermatology/Skin - Other (Mouth sore-lower lip)*3 (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL:: Gastrointestinal - Other (Emesis)*3 (Gastrointestinal disorders) | 1 (1) | 1 (1)
GASTROINTESTINAL:: Gastrointestinal - Other (Erythema mucosa-under tongue & hard palate )*3 (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL:: Gastrointestinal - Other (Gastroesophageal reflux disease)*3 (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL:: Gastrointestinal - Other (Partial bowel obstruction)*3 (Gastrointestinal disorders) | 0 (0) | 1 (1)
PAIN:: Pain - Other (Right inguinal pain)*3 (General disorders) | 0 (0) | 1 (1)
PAIN:: Pain - Other (Rt. thigh pain)*3 (General disorders) | 0 (0) | 1 (2)
PAIN:: Pain - Other (Sternum pain)*3 (General disorders) | 0 (0) | 1 (1)
PAIN:: Pain - Other (Rt. flank)*3 (General disorders) | 1 (1) | 0 (0)
PAIN:: Pain - Other (Rt. ear)*3 (General disorders) | 1 (1) | 0 (0)
PAIN:: Pain - Other (Pain from inserted biliary stents)*3 (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-06-29): https://cdn.clinicaltrials.gov/large-docs/13/NCT00088413/Prot_SAP_ICF_000.pdf